CLINICAL TRIAL: NCT03372421
Title: The Use of Social Stories to Reduce Negative Affect and Improve Satisfaction in Adults Attending an Assessment for Autism Spectrum Disorder
Brief Title: The Use of Social Stories to Reduce Negative Affect and Improve Satisfaction in Adults Attending an ASD Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Richard Jenkinson, Trainee Clinical Psychologist, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: rjenkinson001
Record Dates: First submitted 2017-12-04; First posted 2017-12-13 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be told whether they are in the experimental or control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Story (Experimental): Participants will read information about what to expect from the assessment in the format of a Social Story
  Interventions: Other: Social Story
- Standard Information (Active Comparator): Participants will read standard information about what to expect from the assessment.
  Interventions: Other: Standard Information

INTERVENTIONS:
Other: Social Story — A short story written in the third person about what it's like to attend an assessment for ASD.
  Arms: Social Story
Other: Standard Information — Information the host site currently sends out to patients informing them about what to expect from the assessment
  Arms: Standard Information

SUMMARY:
Many people with Autism Spectrum Disorder (ASD) find the unpredictability of social situations emotionally distressing. It is likely that attending a diagnostic assessment is no exception. Social Stories are short stories that describe a social situation so that people know what to expect. They are written in a way that is accessible to people with ASD. This study will explore whether a Social Story written about a diagnostic assessment can reduce the associated emotional distress and increase people's satisfaction with the process. If so, they could be a simple way that services can better cater for their clients' needs.

DETAILED DESCRIPTION:
An invitation to participate in the study will be included with every appointment letter sent out by the host site(s) whilst recruitment is active. The invitation will invite participants to visit a website (hosted by Qualtrics) where they will be provided with information about the study and asked if they would like to provide informed consent to participate. If consent is given, they will be asked to complete an online version of the Positive and Negative Affect Schedule (PANAS; time 1). Contact information will also be requested at this point.

Participants will then be randomly allocated to either an experimental group or to a control group. Participants in the experimental group will read a Social Story about what to expect from their assessment; participants in the control group will read the standard information the host service sends out about what to expect from their assessment. Participants will be blinded to which group they are in.

If the participants choose to supply a mobile telephone number and email address, an SMS text message and/or email reminder will be sent out one week prior to their assessment and again on the morning of the assessment. These reminders will include hyperlinks to the information about what to expect and will remind them to complete the PANAS once they arrive at their appointment.

On arrival at their assessment (time 2), participants will complete a paper copy of the PANAS questionnaire and will be asked for demographic information. Participants will also be asked to rate the extent that the information they read prior to attending the assessment has helped them to know what to expect thus far. Paper copies of the questionnaire will be left in the waiting area with instructions to hand them into staff once complete.

One week following their assessment (time 3), participants will receive another SMS/email which will include a hyperlink to a post-assessment survey that will ask participants to rate their satisfaction with the assessment and whether they received a diagnosis of ASD. Participants who do not complete this questionnaire after one week will be contacted one final time. All participants will be sent a debriefing sheet.

Hypotheses

1. Compared with participants who read standard, non-social information prior to attending an assessment for ASD, participants who read a Social Story will report, on average, less of an increase in negative affect when attending their assessment, as measured by the negative subscale of the PANAS.
2. Participants who read a Social Story prior to attending an assessment for ASD will report, on average, higher satisfaction (measured via a 5 point Likert scale) with the assessment than participants who read standard, non-social information.
3. Compared with participants who read standard, non-social information prior to attending an assessment for ASD, participants who read a Social Story will report, on average, that the assessment was more predictable (measured via a 5 point Likert scale).

Data Analysis

1. Comparison of means using a 2 (group; SS, control) X 2 (time; time 1, time 2) mixed ANOVA (repeated measures on the time factor). Dependent variable = PANAS score.

   Comparison of means using an independent t-test at time 2. Independent variable = group (2 levels; SS and control). Dependent variable = PANAS score.

   Descriptive statistics.
2. Comparison of means using the Mann-Whitney U test at time 3. Independent variable = group (2 levels; SS and control). Dependent variable = satisfaction score.

   Descriptive statistics.
3. Descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* People who are awaiting an ASD assessment at the host site.
* People who have never visited the site before.

Exclusion Criteria:

* People who do not receive a diagnosis of ASD following the study will not be included in the inferential statistical analysis. However, they will still be participants in the study and their data will be reported descriptively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-05-26 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Affect Schedule | Change scores: baseline and 3 weeks
  A widely used self-report measure of positive and negative affect with good psychometric properties (Crawford & Henry, 2004) and has been used in previous research to measure negative affect in people with ASD (Samson, Huber, & Gross, 2012).

SECONDARY OUTCOMES:
Assessment Satisfaction | 3 weeks
  Participants will be asked to rate their overall satisfaction with the diagnostic assessment, on a 5 point Likert scale.
Predictability | 3 weeks
  Participants will be asked to rate, on a 5 point Likert scale, to what extent the information they read prior to their assessment has thus far helped them to know what to expect from the assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Richard p Jenkinson, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Adult Autism and Neurodevelopmental Service, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared in order to protect the participants' confidentiality

REFERENCES:
- See also: The website of the author of Social Stories with guidance on writing Social Stories. — https://carolgraysocialstories.com/